CLINICAL TRIAL: NCT05460910
Title: Effects of Core Stability Exercises With and Without Treadmill Training on Balance in Children With Down Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0712
Record Dates: First submitted 2022-07-14; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Down Syndrome
Keywords: core stability exercises; balance; treadmill
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- core stability exercise, treadmill (Experimental): core stability exercises and treadmill training
  Interventions: Other: core stability exercises with treadmill
- core stability exercises (Experimental): core stability exercises without treadmill training
  Interventions: Other: core stability exercise without treadmill

INTERVENTIONS:
Other: core stability exercises with treadmill — swiss ball use patient is lying in supine position with 15 repitations and 3 sets.
  Arms: core stability exercise, treadmill
Other: core stability exercise without treadmill — technique used to improve stability
  Arms: core stability exercises

SUMMARY:
To find the effects of core stability exercises with and without treadmill training on balance in children with down syndrome

ELIGIBILITY:
Inclusion Criteria:

* able to stand and walk independently
* able to understand and follow a verbal command
* cutoff score less than 6 or 7 in functional balance in indicated

Exclusion Criteria:

* patients have any neurological issue,
* Instability of atlantoaxial joint
* Vision and hearing loss
* History of fall

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
Berg balance scale | 8th week
  berg balance scale was used to measure the functional balance in children.

SECONDARY OUTCOMES:
Reach test | 8week
  reach test is used to measure the stability in children

CONTACTS AND LOCATIONS:
Overall Officials: Wajiha Shahid, PhD, Principal Investigator — Riphah International University
Locations (1):
- International Therapy Services Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szafraniec R, Baranska J, Kuczynski M. Acute effects of core stability exercises on balance control. Acta Bioeng Biomech. 2018;20(4):145-151. PMID 30520448
- [Background] Alsakhawi RS, Elshafey MA. Effect of Core Stability Exercises and Treadmill Training on Balance in Children with Down Syndrome: Randomized Controlled Trial. Adv Ther. 2019 Sep;36(9):2364-2373. doi: 10.1007/s12325-019-01024-2. Epub 2019 Jul 12. PMID 31301057
- [Background] Amini HA, Fazel Kalkhoran J, Salehi M, Jazini F. Effect of backward walking training on improves postural stability in children with down syndrome. International Journal of Pediatrics. 2016;4(7):2171-81.